CLINICAL TRIAL: NCT05771467
Title: Evaluation of Retinal Microvascular Change That May Develop in After Open Globe Injury With Optical Coherence Tomography
Brief Title: Evaluation of Retinal Microvascular Change That May Develop in After Open Globe Injury
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Aslı Çetinkaya Yaprak, Associate Professor, Akdeniz University
Other Study IDs: AKDENIZ-GOZ-001
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Eye Injury Trauma
Keywords: Eye Injury Trauma; Open Globe Injury; Optical Coherence Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma Group: Non-trauma eye after open globe injury determine retinal microvascular changes
  Interventions: Diagnostic Test: Comprehensive Ophthalmologic Examination
- Control Group: Investigation of retinal microvascular circulation in age- and sex-matched healthy volunteers
  Interventions: Diagnostic Test: Comprehensive Ophthalmologic Examination

INTERVENTIONS:
Diagnostic Test: Comprehensive Ophthalmologic Examination — Measurements of best-corrected visual acuity, refractive error, intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination, and anterior segment parameters, optical coherence tomography angiography (OCTA)
  Other Names: Optical Coherence Tomography Angiography (OCTA); Biometry; Auto refractometry; Non contact tonometry

SUMMARY:
The aim of this study is to evaluate posterior segment changes in the non-traumatic eye after open globe injury.

DETAILED DESCRIPTION:
Globe injuries can be classified as either closed- or open-globe injuries, based on the integrity of the sclera and cornea. Open-globe injury (OGI) is characterized by a full-thickness wound of the ocular wall.

As one of the most severe forms of ocular trauma, open-globe injury (OGI) causes significant vision loss. Timely and meticulous repair of these injuries can improve patient outcomes.

OGI by rupture often occurs at the weakest point of the eye wall, which may or may not be at the actual injury site. The rupture site is most commonly found in the sclera concentric to the limbus, just posterior to the insertion of the extraocular muscles.

After trauma, changes may occur in the non-trauma eye. Retinal and choroidal circulation may change as a result of adaptation mechanisms. In this study, we evaluated the vascular densities of the control group and post-traumatic non-trauma eye.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Unilateral eye injury

Exclusion Criteria:

* Be under the age of 18
* Usage of systemic drugs or topical ocular drops
* Bilateral eye injury
* Having systemic disease, having ocular pathology that may decrease visual acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle age, predominantly male
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Samet Atlıhan, MD, 1, Principal Investigator — Akdeniz University Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Aslı Çentinkaya Yaprak, Antalya
  - Yusuf Samet Atlıhan, Antalya

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Trauma Group: Non-Trauma Eye After Open-Globe Injury All subjects underwent a comprehensive ophthalmologic examination, which included refractive error (Nidek ARK-700A, Nidek Co., Ltd, Gamagori, Japan), best corrected visual acuity (BCVA), IOP/Fully Automatic Tonometer, NIDEK NT-2000, Nidek Co., Ltd., Aichi, Japan), biometry and axial length (AL) (IOLMASTER 500, Carl Zeiss Meditec AG, Jena, Germany), slit-lamp examination of the anterior and posterior segments, Scheimflug Topography (Pentecam Oculus Optikgeräte GmbH, Wetzlar, Germany), and retinal and choroidal thickness and microvascular circulation of the retina and choroid were measured and recorded with Swept-Source Optical Coherence Tomography Angio™ (Topcon Corp, Japan). The BCVA was converted into the logarithm of minimal angle resolution (logMAR). Of the individuals included in the study, anterior chamber depth (ACD), anterior chamber volume (ACV), thinnest corneal thickness (TCT), astigmatism value (AST), corneal volume (CV), axial length (AL), spherical equivalent (SFEQ), intraocular lens power (ILP), VA (visual acuity), central retinal thicness (CRT), central choroidal thickness (CCT), superficial retinal circulation (SRC), deep retinal circulation (DRC) and choriocapillaris circulation (CC) data were recorded. The patients were followed for approximately six months, examined at one week, one month and three months after the trauma, and a total of three measurements were taken from the subjects.
- Control Group: Age-, sex-matched healthy volunteers
  All subjects underwent a comprehensive ophthalmologic examination, which included refractive error (Nidek ARK-700A, Nidek Co., Ltd, Gamagori, Japan), best corrected visual acuity (BCVA), IOP/Fully Automatic Tonometer, NIDEK NT-2000, Nidek Co., Ltd., Aichi, Japan), biometry and axial length (AL) (IOLMASTER 500, Carl Zeiss Meditec AG, Jena, Germany), slit-lamp examination of the anterior and posterior segments, Scheimflug Topography (Pentecam Oculus Optikgeräte GmbH, Wetzlar, Germany), and retinal and choroidal thickness and microvascular circulation of the retina and choroid were measured and recorded with Swept-Source Optical Coherence Tomography Angio™ (Topcon Corp, Japan). The BCVA was converted into the logarithm of minimal angle resolution (logMAR). Of the individuals included in the study, anterior chamber depth (ACD), anterior chamber volume (ACV), thinnest corneal thickness (TCT), astigmatism value (AST), corneal volume (CV), axial length (AL), spherical equivalent (SFEQ), intraocular lens power (ILP), VA (visual acuity), central retinal thicness (CRT), central choroidal thickness (CCT), superficial retinal circulation (SRC), deep retinal circulation (DRC) and choriocapillaris circulation (CC) data were recorded.
Period: Overall Study
Arm/Group | Trauma Group | Control Group
Started | 50 | 50
Completed | 44 | 47
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 6 | 3

BASELINE CHARACTERISTICS:
Population: older 18 years
Groups:
- Trauma Group: Non-Trauma Eye After Open-Globe Injury
  Optical Coherence Tomography Angiography (OCTA) • Biometry • Auto refractometry • Non contact tonometry: Ophthalmologic Examination Measurements of best-corrected visual acuity, refractive error, intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination, and anterior segment parameters, optical coherence tomography angiography (OCTA)
- Control Group: Age-, sex-matched healthy volunteers
  Optical Coherence Tomography Angiography (OCTA) • Biometry • Auto refractometry • Non contact tonometry: Ophthalmologic Examination Measurements of best-corrected visual acuity, refractive error, intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination, and anterior segment parameters, optical coherence tomography angiography (OCTA)
- Total: Total of all reporting groups
Arm/Group | Trauma Group | Control Group | Total
Number analyzed (Participants) | 44 | 47 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 36 | 71
  >=65 years | 9 | 11 | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 51 (20.6) | 43 (17.5) | 44 (19.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 23 | 29 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 44 | 47 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 44 | 47 | 91

OUTCOME MEASURES:

1. Primary Outcome: Corneal Thickness
Description: Corneal thickness in mikrometer value
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Total Group: Total number of cases
Arm/Group | Trauma Group | Control Group | Total Group
Number analyzed (Participants) | 44 | 47 | 91
microns | 542.23 (27.47) | 546.16 (46.03) | 544.32 (35.3)

2. Primary Outcome: Anterior Chamber Volume
Description: Anterior chamber volume in mm3
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: Cubic micrometre
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
Cubic micrometre | 177.97 (28.46) | 165.9 (26.73)

3. Primary Outcome: Anterior Chamber Depth
Description: Anterior chamber depth in mm
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
milimeters | 2.93 (0.25) | 3.05 (0.29)

4. Primary Outcome: Anterior Chamber Angle
Description: Anterior chamber angle in degree
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
degree | 38.87 (6.42) | 37.8 (4.74)

5. Primary Outcome: Lens Power
Description: in diopters
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
diopters | 20.98 (0.35) | 20.26 (0.44)

6. Primary Outcome: Steep Keratometry
Description: in Diopters measured with pentacam
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
diopters | 44.22 (1.64) | 44.57 (1.82)

7. Primary Outcome: Tonometry
Description: Intraocular pressure measurement in mmHg
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: milimeter mercury
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
milimeter mercury | 14.74 (0.49) | 15.78 (0.35)

8. Primary Outcome: Axial Length
Description: Axial length in mm
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
milimeters | 23.86 (0.94) | 23.36 (0.72)

9. Primary Outcome: Optic Nerve Head Vessel Density
Description: Optic nerve head vessel density assessed with optical coherence tomography angiography
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: vessels/mm^2
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
vessels/mm^2 | 23.22 (5.2) | 25.2 (4.4)

10. Primary Outcome: Choriocapillaris Flow Area
Description: Choriocapillaris flow area assessed with optical coherence tomography angiography
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
mm^2 | 36.88 (1.52) | 36.53 (1.89)

11. Primary Outcome: Subfoveal Central Macular Thickness
Description: Subfoveal central macular thickness assessed with optical coherence tomography
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Trauma Group | Control Group
Number analyzed (Participants) | 44 | 47
microns | 321.42 (24.52) | 311.57 (31.13)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Trauma Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT05771467/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/67/NCT05771467/ICF_001.pdf